CLINICAL TRIAL: NCT02915432
Title: A Multi-Center, Open Label Phase Ib/II Clinical Study to Evaluate JS001 in Patients With Advanced Gastric Adenocarcinoma, Esophageal Squamous Cell Carcinoma, Nasopharyngeal Carcinoma and Head and Neck Squamous Cell Carcinoma
Brief Title: The Study to Evaluate Toripalimab (JS001) in Patients With Advanced GC, ESCC, NPC, HNSCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JS001-Ib-CRP-1.0
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Gastric Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Nasopharyngeal Carcinoma; Head and Neck Squamous Cell Carcinoma
Keywords: Anti PD-1; JS001; Gastric Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Nasopharyngeal Carcinoma; Head and Neck Squamous Cell Carcinoma; Simon's Two Stage; ORR
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Nasopharyngeal Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 mg/kg anti-PD-1 mAb JS001 Q2W (Experimental): Subjects will be eligible for this study after they fulfill the inclusion criteria and exclusion criteria. Subjects diagnosed as the gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, or head and neck squamous cell carcinoma will receive treatment at the dose of 3 mg/kg.
  Interventions: Biological: 3 mg/kg anti-PD-1 mAb JS001 Q2W
- 360 mg anti-PD-1 mAb JS001 Q3W (Experimental): Subjects will receive corresponding regimen of standard first-line chemotherapy combined with JS001 360 mg once every 3 weeks (Q3W). JS001 360 mg Q3W can be administrated after the end of chemotherapy until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, and withdrawal of informed consent by the subject, or death.
  Interventions: Biological: 360 mg anti-PD-1 mAb JS001 Q3W
- 240mg anti-PD-1 mAb JS001 Q3W (Experimental): Subjects will receive corresponding regimen of standard first-line chemotherapy combined with JS001 240 mg once every 3 weeks (Q3W). JS001 240 mg Q3W can be administrated after the end of chemotherapy until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, and withdrawal of informed consent by the subject, or death
  Interventions: Biological: 240mg anti-PD-1 mAb JS001 Q3W

INTERVENTIONS:
Biological: 3 mg/kg anti-PD-1 mAb JS001 Q2W — This study is planned to conduct the 3 mg/kg dose group study at first. After enrollment, the subjects will be administered every 2 weeks (Q2W) with 4 weeks as a cycle, until absence of further benefits, acceptable toxicity, investigator decision, consent withdrawal or death.
  If patient experiences 1st onset of disease progression and investigator judges that patient will obtain clinical benefit from the study treatment, patient can continue the study treatment after the discussion between investigator and medical monitor from sponsor or authorized CRO and approval is obtained afterwards. If the subject develops 2nd disease progression after 1st disease progression, he/she should permanently withdraw from the study treatment.
  Other Names: toripalimab, TAB001
  Arms: 3 mg/kg anti-PD-1 mAb JS001 Q2W
Biological: 360 mg anti-PD-1 mAb JS001 Q3W — Subjects will receive corresponding regimen of standard first-line chemotherapy combined with JS001 360 mg once every 3 weeks (Q3W). JS001 360 mg Q3W can be administrated after the end of chemotherapy until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, and withdrawal of informed consent by the subject, or death.
  Other Names: toripalimab, TAB001
  Arms: 360 mg anti-PD-1 mAb JS001 Q3W
Biological: 240mg anti-PD-1 mAb JS001 Q3W — Subjects will receive corresponding regimen of standard first-line chemotherapy combined with JS001 240 mg once every 3 weeks (Q3W). JS001 240 mg Q3W can be administrated after the end of chemotherapy until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, and withdrawal of informed consent by the subject, or death.
  Other Names: toripalimab, TAB001
  Arms: 240mg anti-PD-1 mAb JS001 Q3W

SUMMARY:
The purpose of this study is to preliminarily evaluate anti-tumor activity of a Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Infusion (JS001) in treating advanced gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma and head and neck squamous cell carcinoma and to determine the recommended phase II dose (RP2D)

DETAILED DESCRIPTION:
Overall Design:

This is a multicenter, open-label, phase Ib/II clinical study of Toripalimab Injection (JS001) in patients with gastric adenocarcinoma (GC), esophageal squamous cell carcinoma (ESCC), nasopharyngeal carcinoma (NPC), or head and neck squamous cell carcinoma (HNSCC). On the basis of the results of safety and pharmacokinetic data in the phase I study of JS001, 3 mg/kg is determined as the recommended dose of the 2-week monotherapy regimen, and no study on the 10 mg/kg cohorts will be conducted any more. And the corresponding 240 mg and 360 mg are determined as the corresponding exploratory doses of the 3-week combined treatment regimens.

Eligible subjects will be selected based on the inclusion and exclusion criteria: subjects with gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, or head and neck squamous cell carcinoma (cohort 1, 2, 3, 4, respectively) will receive treatment at the dose of 3 mg/kg. While subjects with advanced gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, or head and neck squamous cell carcinoma (cohort 5, 6, 7, 8, respectively), who have not received any treatment before, will be treated with the corresponding 3-week regimen of standard first-line chemotherapy combined with JS001 240 mg or 360 mg .

Study Treatment:

The study on the 3 mg/kg cohorts is planned to be conducted first in cohort 1, 2, 3, 4 in this trial. After enrollment, the subjects will receive study treatment once every 2 weeks (Q2W) with 4 weeks as a cycle, until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, withdrawal of informed consent by the subject, or death.

The study of cohort 5, 6, 7, and 8 will be carried out in the sites designated by the sponsor. Subjects will receive corresponding regimen of standard first-line chemotherapy combined with JS001 240 mg or 360 mg once every 3 weeks (Q3W) (see Section 3.1 Overall Design for details). JS001 240 mg or 360 mg Q3W can be administrated after the end of chemotherapy until absence of further benefits judged by the investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, and withdrawal of informed consent by the subject, or death.

If the subject experiences disease progression but the subject can still obtain clinical benefit from the study treatment of JS001 according to the investigator, the subject can continue the study treatment if an approval is obtained after discussion between the investigator and the medical monitor from the sponsor or the authorized CRO. If the subject develops disease progression for a second time, he/she should permanently withdraw from the study treatment.

Tumor Assessment:

During the study, for cohort 1, 2, 3, and 4, tumor responses will be evaluated every 8 weeks in the first year according to RECIST 1.1, and every 12 weeks thereafter. Tumor responses will also be evaluated according to irRECIST at the same frequency with that conducted according to RECIST 1.1 until disease progression, death or loss of follow up (whichever comes first). For cohort 5, 6, 7, and 8, tumor responses will be evaluated every 6 weeks (± 3 days) in the first year according to RECIST 1.1 and irRECIST, and every 12 weeks thereafter until disease progression, death or loss of follow up (whichever comes first).

The radiographic data of the subjects will be collected for review by IRC. The IRC will evaluate the corresponding study endpoints based on tumor responses, but no such evaluation is planned for cohort 5, 6, 7 and 8.

Pharmacokinetics:

At least 10 of the subjects (no requirements on indications) in JS001 3 mg/kg cohorts at the sponsor-designated study sites should complete the pharmacokinetic blood sampling in the first 3 cycles of study treatment until 60 days after the end of study treatment. If a subject did not complete the scheduled sample collection in the first 3 cycles of study treatment due to any reason, another subject should be added.

Corresponding pharmacokinetic blood samplings will also be conducted for cohort 5, 6, 7, and 8, to evaluate the pharmacokinetic characteristics of JS001 used in the combined treatment with chemotherapy. At least 3 patients will be selected for blood sampling in each cohort.

Acquisition of Tumor Tissue Specimens:

Subjects with esophageal squamous cell carcinoma, gastric adenocarcinoma (including adenocarcinoma at esophageal-gastric conjunction), nasopharyngeal carcinoma, or head and neck squamous cell carcinoma must provide acceptable tumor tissue specimens (fresh tumor tissue specimens for biopsy before enrollment are preferred) prior to enrollment for future use in subsequent exploratory studies.

Any subject with the response confirmed as partial response (PR) and/or progressive disease (PD) is encouraged to voluntarily participate in the selectable biomarkers study if tumor tissues can be obtained from him/her. And in the selectable biomarkers study, they will provide tumor tissues for exploratory study on the correlation between tumor markers and the level of anti-tumor responses.

All the tumor tissue specimens provided will be sent to the designated central laboratory for evaluation.

End of Study:

The primary endpoint of the study is ORR. The study will be completed at 12 months after the last patient in and data analysis will be conducted then. If by that time there are still some subjects receiving study treatment, these subjects will be transferred to an extension study to continue the study treatment until absence of further benefits judged by investigator, disease progression, occurrence of intolerable toxicity, investigator's decision, withdrawal of informed consent by subject, or death.

ELIGIBILITY:
"Inclusion Criteria Subjects may be entered in the study only if they meet all of the following criteria:

1. Fully understand the study and signed the Informed Consent Form (ICF) voluntarily;
2. Subjects with histologically and/or cytologically confirmed advanced and/or metastatic gastric adenocarcinoma (including adenocarcinoma at esophageal-gastric conjunction), esophageal squamous cell carcinoma, nasopharyngeal carcinoma, or head and neck squamous cell carcinoma, who meet the following conditions (not applicable to cohort 5, 6, 7, and 8):

   Subjects with gastric adenocarcinoma must have received at least one line of anti-tumor treatment for advanced gastric adenocarcinoma and have documented tumor progression or be intolerable to the current available chemotherapy regimen. Subjects who have recurrence or metastasis within 6 months after completion of concomitant adjuvant or neoadjuvant chemotherapy of radical operation are eligible to this study; Subjects with esophageal squamous cell carcinoma must have received at least one line of treatment for advanced esophageal squamous cell carcinoma (including but not limited to anticancer drug treatment or radio-chemotherapy) and have documented tumor progression or be intolerable to the current chemotherapy regimen. Subjects who have recurrence or metastasis within 6 months after completion of concomitant adjuvant or neoadjuvant therapy (including but not limited to chemotherapy or radio-chemotherapy) of radical operation are eligible to this study;

   Subjects with nasopharyngeal carcinoma or head and neck squamous cell carcinoma who have received at least one line of treatment for advanced nasopharyngeal carcinoma or head and neck squamous cell carcinoma (including but not limited to anticancer drug treatment or radio-chemotherapy) and have documented tumor progression or be intolerable to other current chemotherapy regimens. Subjects with recurrence or metastasis within 6 months after completion of concomitant adjuvant or neoadjuvant radio-chemotherapy of radical operation are eligible to this study (only applies for Version 4.1 and the previous ones); while for the working protocol version 5.0, subjects with nasopharyngeal carcinoma can be enrolled only if they meet the following criteria:

   subjects having received at least two lines of treatment for advanced nasopharyngeal carcinoma (including but not limited to anticancer drug treatment and radio-chemotherapy), who are confirmed to have tumor progression or be intolerable to other current chemotherapy regimens; adjuvant or neoadjuvant radio-chemotherapy after radical surgery can be considered as one line of treatment if tumor recurrence or metastasis occurred within 6 months after the end of the radio-chemotherapy.
3. At least one measurable lesion (according to RECIST 1.1); Note: Any lesion which received radiotherapy treatment previously cannot be regarded as a target lesion, unless that it has definitely progressed after radiotherapy.
4. Agree to provide archived tumor tissue specimens or have biopsy to collect tumor tissues for PD-L1 IHC measurement in the central laboratory;
5. Males or females aged between 18 and 75 years old;
6. ECOG score of 0-1;
7. Life expectancy ≥ 3 months;
8. The results of laboratory tests performed within 7 days prior to enrollment must meet the following criteria:

   1. Neutrophils ≥ 1.5×109/L (not applicable to cohort 5, 6, 7, and 8);
   2. Platelets ≥ 75×109/L (not applicable to cohort 5, 6, 7, and 8);
   3. Hemoglobin ≥ 90 g/L (without receiving infusion of concentrated red blood cells within 2 weeks);
   4. Serum creatinine ≤ 1.5× upper limit of normal (ULN), or creatinine clearance > 50 mL/min (not applicable to cohort 5, 6, 7, and 8);
   5. Serum total bilirubin ≤ 1.5×ULN (total bilirubin ≤ 3×ULN are acceptable for subjects with Gilbert syndrome);
   6. Both AST and ALT ≤ 2.5×ULN; ALT and AST ≤ 5×ULN are acceptable for subjects with liver metastasis;
9. Serum pregnancy test result must be confirmed as negative for women of childbearing potential within 28 days prior to enrollment and the subjects must agree to take effective contraception measures throughout the study treatment period until 60 days after the end of study treatment. Women of childbearing potential are defined as women with sexual maturity, who meet any of the following conditions: 1) no hysterectomy or bilateral oophorectomy; 2) without natural menopause for a consecutive 24 months (patients with menopause after cancer treatment may also have childbearing potential) (i.e. menstruation occurred at any time during the previous consecutive 24 months) (not applicable to cohort 5, 6, 7, and 8).

Female partners of childbearing potential of the male subjects should also follow the contraception requirements.

Other special inclusion criteria for cohort 5, 6, 7, and 8.

1. Subjects with histologically and/or cytologically confirmed advanced and/or metastatic gastric adenocarcinoma (including adenocarcinoma at esophageal-gastric conjunction), esophageal squamous cell carcinoma, nasopharyngeal carcinoma, or head and neck squamous cell carcinoma, who meet any of the following conditions:

   1. Subjects who have not received any systematic treatment.
   2. Subjects who have received any neoadjuvant chemotherapy, adjuvant chemotherapy for the purpose of curing must experience a period for at least 6 months from the end of the last chemotherapy to tumor progression.
   3. Subjects with head and neck squamous cell carcinoma must have received radiotherapy for the purpose of curing, and the period from the end of radiotherapy to tumor progression must be at least 1 year.
   4. For subjects with gastric carcinoma, Her2 negative is required. HER2 positive is defined as IHC 3+ or IHC 2+ combined with ISH+, and ISH positive is defined as the ratio of the number of HER2 gene copies to the number of CEP17 signals ≥ 2.0.
2. Results of laboratory test conducted within 7 days before enrollment must meet the following criteria:

   1. Neutrophils ≥ 2×109/L; WBC count ≥ 4×109L and < 15×109/L
   2. Platelets ≥ 100×109/L;
   3. Hemoglobin ≥ 90 g/L (no infusion of concentrated red blood cells within 2 weeks);
   4. Creatinine clearance rate > 60 mL/min, based on the predicted value of Cockcroft-Gault glomerular filtration rate:

      (140 - age) × (weight, kg) × (0.85, if females) 72× (serum creatinine, mg/dL) Or: (140 - age) × (weight, kg) × (0.85, if females) 0.818 × (serum creatinine, μmol/L)
   5. Serum total bilirubin ≤ 1.5 × ULN (total bilirubin ≤ 3 × ULN are acceptable for subjects with Gilbert syndrome);
   6. INR and aPTT ≤ 1.5 × ULN, applies only to subjects who have not received anticoagulation; and for subjects who are receiving anticoagulation, the dose for anticoagulation must be stable.
3. Serum pregnancy test result must be confirmed as negative for women of childbearing potential within 28 days prior to enrollment and the subjects must agree to take effective contraception measures throughout the study treatment period until 6 months after the end of chemotherapy or 60 days after the end of study treatment (whichever comes last). Women of childbearing potential are defined as women with sexual maturities, who meet any of the following conditions: 1) no hysterectomy or bilateral oophorectomy; 2) without natural menopause for a consecutive 24 months (patients with menopause after cancer treatment may also have childbearing potential) (i.e. menstruation occurred at any time during the previous consecutive 24 months) .

Female partners of childbearing potential of the male subjects should also follow the contraception requirements.

Subjects fulfilling any of the following conditions cannot be enrolled in the study:

1. Known hypersensitivity to citric acid monohydrate, dihydrate sodium citrate, mannitol or polysorbate (components of the investigational drug);
2. Anti-tumor treatment with cytotoxic drugs, biological drugs (e.g. monoclonal antibody), immunotherapy (e.g. interleukin 2 or interferon), or other investigational drugs within 4 weeks prior to enrollment;
3. Tyrosine kinase inhibitor treatment within 2 weeks prior to enrollment;
4. Radiotherapy within 4 weeks prior to enrollment, or radioactive drugs within 8 weeks prior to enrollment. However, patients receiving local palliative radiotherapy for bone metastasis lesions can be included;
5. Subjects with any major surgical operation within 4 weeks prior to enrollment or who have not completely recovered from the prior operation (for the definition of major surgical operation, please refer to the Level 3 and Level 4 operations stipulated in the Management of Clinical Application of Medical Technology enforced on May 1, 2009);
6. Toxicity due to any previous anticancer treatment has not recovered to CTCAE Grade 0-1, excluding the following conditions:

   1. Alopecia;
   2. Pigmentation;
   3. Peripheral nerve toxicity recovered to < CTCAE Grade 2 (not applicable to cohort 5, 6, 7, and 8, subjects are not eligible if peripheral neurotoxicity does not restore to normal);
   4. Long-term toxicity related to radiotherapy, which will not fully recover as judged by the investigator.
7. Central nervous system metastasis with clinical symptoms (e.g. brain edema, hormone intervention required, or progression of brain metastasis) and/or carcinomatous meningitis. Subjects with prior treatment for brain or meningeal metastasis can be included if they have remained stable clinically for at least 2 months and systemic hormone treatment (Prednisone at a dose of > 10 mg/day or other equivalent hormone formulations) has been discontinued for more than 4 weeks;
8. Subjects with nasopharyngeal carcinoma or head and neck squamous cell carcinoma, who are found to have necrotic lesions by examination within 4 weeks prior to enrollment, for which there is a potential risk of massive hemorrhage as judged by the investigator;
9. Previous or other concurrent malignant tumors (expect for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervix carcinoma in situ, and other malignant tumors which were effectively controlled without treatment over the past 5 years);
10. Any active autoimmune disease or history of any autoimmune disease (including but are not limited to interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism or hypothyroidism. Patients with vitiligo or asthma (in childhood) which was completely resolved and without need of any intervention in adulthood can be included. However, subjects with asthma which needs bronchodilator for medical intervention cannot be included);
11. Previous treatments with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody which acts on T-cell co-stimulatory or checkpoint pathway);
12. Subjects diagnosed with active tuberculosis (TB), who are receiving anti-tuberculosis therapy or used to have anti-tuberculosis therapy within 1 year prior to screening;
13. Concomitant diseases requiring long-term treatment with immunosuppressive drugs, or corticosteroids at an effective immunosuppressive dose (Prednisone at a dose of > 10 mg/day or other equivalent hormone formulations) for systemic or local treatment purpose;
14. Subjects who have received any anti-infection vaccine (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment;
15. Pregnant or lactating women
16. Positive test for HIV;
17. Positive test for HBsAg, with HBV DNA copies detected as positive (quantitative measurements ≥ 1000 cps/mL);
18. Positive test for chronic Hepatitis C in blood screening test (HCV antibody positive); Any other clinical significant disease or condition, which as evaluated by the investigator, may affect the protocol compliance, signing of inform consent form (ICF), or not suitable to participate into this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 1.5 approximately years
  To preliminarily evaluate the anti-tumor activity of Toripalimab Injection (former name: Recombinant humanized anti-PD-1 monoclonal antibody for injection, JS001) in treating advanced gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma, and head and neck squamous cell carcinoma.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 1.5 approximately years
Disease control rate (DCR) | Up to 1.5 approximately years
Progression free survival (PFS) | Up to 1.5 approximately years
Overall survival (OS) | Up to 1.5 approximately years
afety: incidence and severity of adverse events, and clinically significant laboratory abnormalities | Up to 1.5 approximately years
The frequencies of positive and negative anti-drug antibody (ADA) test compared with baseline | Up to 1.5 approximately years
Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) | Up to 1.5 approximately years
Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years
Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years
t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb | Up to 1.5 approximately years
Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years
Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years
Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb | Up to 1.5 approximately years

OTHER OUTCOMES:
Correlation between PD-L1 expression in tumor tissue and the anti-tumor activity of JS001 demonstrated in the analysis | Up to 1.5 approximately years
Correlation between EBV expression in tumor tissue of esophageal squamous cell carcinoma and gastric adenocarcinoma and the anti-tumor activity of JS001 demonstrated in the analysis | Up to 1.5 approximately years
Correlation between EBV expression in tumor tissue and blood of nasopharyngeal carcinoma and the anti-tumor activity of JS001 demonstrated in the analysis | Up to 1.5 approximately years
Correlation between HPV expression in tumor tissue of head and neck squamous cell carcinoma and the anti-tumor activity of JS001 demonstrated in the analysis | Up to 1.5 approximately years
Correlation between MSI expression in tumor tissue of esophageal squamous cell carcinoma and gastric adenocarcinoma and the anti-tumor activity of JS001 demonstrated in the analysis | Up to 1.5 approximately years
Correlation between the expression of other potential pharmacodynamic indexes and the anti-tumor activity of JS001 demonstrated in the analysi | Up to 1.5 approximately years
Correlation of the changes of TBNK lymphocytes subgroup in patients receiving chemotherapy combined with JS001 and its correlation with the anti-tumor activity | Up to 1.5 approximately years

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (23):
- China (23):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army (PLAGH), Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer center, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Tumor Hospital of Hebei Province, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- [Derived] Wei XL, Xu JY, Wang DS, Chen DL, Ren C, Li JN, Wang F, Wang FH, Xu RH. Baseline lesion number as an efficacy predictive and independent prognostic factor and its joint utility with TMB for PD-1 inhibitor treatment in advanced gastric cancer. Ther Adv Med Oncol. 2021 Jan 31;13:1758835921988996. doi: 10.1177/1758835921988996. eCollection 2021. PMID 33613701
- [Derived] Wang FH, Wei XL, Feng J, Li Q, Xu N, Hu XC, Liao W, Jiang Y, Lin XY, Zhang QY, Yuan XL, Huang HX, Chen Y, Dai GH, Shi JH, Shen L, Yang SJ, Shu YQ, Liu YP, Wang W, Wu H, Feng H, Yao S, Xu RH. Efficacy, Safety, and Correlative Biomarkers of Toripalimab in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial (POLARIS-02). J Clin Oncol. 2021 Mar 1;39(7):704-712. doi: 10.1200/JCO.20.02712. Epub 2021 Jan 25. PMID 33492986
- [Derived] Wang F, Wei XL, Wang FH, Xu N, Shen L, Dai GH, Yuan XL, Chen Y, Yang SJ, Shi JH, Hu XC, Lin XY, Zhang QY, Feng JF, Ba Y, Liu YP, Li W, Shu YQ, Jiang Y, Li Q, Wang JW, Wu H, Feng H, Yao S, Xu RH. Safety, efficacy and tumor mutational burden as a biomarker of overall survival benefit in chemo-refractory gastric cancer treated with toripalimab, a PD-1 antibody in phase Ib/II clinical trial NCT02915432. Ann Oncol. 2019 Sep 1;30(9):1479-1486. doi: 10.1093/annonc/mdz197. PMID 31236579